CLINICAL TRIAL: NCT06330012
Title: Spatial Transcriptomic Approach for Revealing the Resistance Mechanism of Trastuzumab Deruxtexan in HER2 Positive Breast Cancer Patients.
Brief Title: The Resistance Mechanism of Trastuzumab Deruxtexan in HER2 Positive Breast Cancer Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JI-YEON, KIM, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GeoMx_Breast
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spatial transcriptomic approch (Experimental): Spatial transcriptomic approch for revealing the resistance mechanism of trastuzumab deruxtexan in HER2 positive breast cancer patients.
  Interventions: Diagnostic Test: GeoMx data analysis with clinical outcome

INTERVENTIONS:
Diagnostic Test: GeoMx data analysis with clinical outcome — 1. List of HER2 positive breast cancer
     * Stage IV disease
     * Treated with T-Dxd
     * Available FFPE samples
  2. Prepare tissue for digital spatial proteomics
     * FFPE/H&E slide
     * Region of Interest(ROI) check
     * Make a Tissue microarray
     * Prepare special slide for GeoMx
  3. GeoMx data analysis with clinical outcome

SUMMARY:
This study is the spatial transcriptomic approach for revealing the resistance mechanism of trastuzumab deruxtexan in HER2 positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive breast cancer
* Stage IV disease
* Treated with T-Dxd
* Available FFPE samples

Exclusion Criteria:

* TNBC breast cancer
* Hormone receptor positive breast cancer
* Non-available FFPE samples
* Treated except T-Dxd

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Spatial transcriptomic analysis | Before chemotherapy, curative surgery
  Protein expression and relationship protein-protein in HER2 positive breast cancer tumor cells and tumor microenvironment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ji-Yeon Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No